CLINICAL TRIAL: NCT06474949
Title: Local Anesthetic for Plateau Fractures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jonah Hebert-Davies, Assistant Professor, School of Medicine: Orthopedics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00017105
Record Dates: First submitted 2024-03-29; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Tibial Plateau Fractures
Keywords: tibial plateau fracture
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient is asleep at time of injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Active Comparator): Bupivacaine
  Interventions: Drug: Bupivacaine injection
- Saline (Placebo Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Bupivacaine injection — Injection at end of Open Reduction Internal Fixation
  Arms: Bupivacaine
Other: Saline — Injection at end of Open Reduction Internal Fixation
  Other Names: Placebo
  Arms: Saline

SUMMARY:
Subjects may receive an injection at the end of the surgery to fix their broken leg that may reduce their pain and hospital stay

DETAILED DESCRIPTION:
Subjects will be randomized to bupivicaine or saline injection in the joint at the end of Open Reduction Internal Fixation of the tibial plateau fracture

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 year ,
* tibial plateau fracture undergoing Open Reduction and fixation"

Exclusion:

* allergy to bupivacaine
* Prolonged external fixator use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain in the knee visual analogue scale 11 point scale 0(no pain) -10 (worst pain) | From date of hospitalization to end of follow-up at 6 months
  Pain at time of visit

SECONDARY OUTCOMES:
Length of stay for hospitalization | From date of hospitalization up to one month post surgery
  Length of stay for hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jonah Hebert-Davies, Principal Investigator — University of Washington

DOCUMENTS (1):
  • Study Protocol (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT06474949/Prot_000.pdf